CLINICAL TRIAL: NCT06014814
Title: Pulsed Field Ablation Under Mild Conscious Sedation - A Feasibility Study
Brief Title: Feasibility of Pulsed Field Ablation Under Mild Conscious Sedation
Status: Completed | Type: Observational
Sponsor: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: PFA-Sedation-Study; IRAS (Other: 320883)
Record Dates: First submitted 2023-07-17; First posted 2023-08-28 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pulsed Field Ablation - General Anaesthesia: Patients undergoing pulsed field ablation for atrial fibrillation under general anaesthetic.
  Interventions: Procedure: Catheter ablation
- Pulsed Field Ablation - Mild Conscious Sedation: Patients undergoing pulsed field ablation for atrial fibrillation under mild conscious sedation.
  Interventions: Procedure: Catheter ablation

INTERVENTIONS:
Procedure: Catheter ablation — Catheter ablation of atrial fibrillation

SUMMARY:
Prospective case-control study comparing pulsed field ablation for atrial fibrillation under mild conscious sedation vs standard of care (general anaesthesia).

DETAILED DESCRIPTION:
This study will prospectively assess 40 patients (20 per arm). Those in the general anaesthesia arm will undergo routine clinical practice. Those in the mild conscious sedation arm will undergo pulsed field ablation with intravenous sedation but without general anaesthesia, though conversion to general anaesthesia is allowed if the patient does not tolerate the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients clinically referred for and undergoing catheter ablation of atrial fibrillation using pulsed field ablation

Exclusion Criteria:

* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been referred clinically for ablation of atrial fibrillation, and will be undergoing this procedure using pulsed field ablation. Patients will not be randomised in this feasibility study - the decision to perform the procedure under mild conscious sedation will be made between the consultant and the patient.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-08-21 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2024-06-11 (Actual)

PRIMARY OUTCOMES:
Number and Percentage of Patients Converting to General Anaesthesia in the Conscious Sedation Arm | Intraprocedural
  Requirement for conversion to general anaesthesia from mild conscious sedation

SECONDARY OUTCOMES:
Patient experience (Pain; Relative) | Intraprocedural
  5 point Likert scale for pain during the procedure, 1 = much worse than expected, 5 = much better than expected
Patient experience (Discomfort; Relative) | Intraprocedural
  5 point Likert scale for discomfort (for example, thumping, heart racing, muscle twitching) during the procedure, 1 = much worse than expected, 5 = much better than expected
Patient experience (Anxiety; Relative) | Intraprocedural
  5 point Likert scale for anxiety during the procedure, 1 = much worse than expected, 5 = much better than expected
Patient experience (Pain; Absolute) | Intraprocedural
  Visual analogue score for pain during the procedure; 1-100, 1 = none, 100 = worst imaginable
Patient experience (Discomfort; Absolute) | Intraprocedural
  Visual analogue score for discomfort (for example thumping, heart racing, muscle twitching) during the procedure (1-100, 1 = none, 100 = worst imaginable)
Patient experience (Anxiety; Absolute) | Intraprocedural
  Visual analogue score anxiety during the procedure; 1-100, 1 = none, 100 = worst imaginable
Post-operative discomfort (Visual analogue score) | Immediately after the procedure
  Visual analogue scores for sites post-operative discomfort (groin, chest, throat), (1-100, 1 = none, 100 = worst imaginable)
Friends and family test | Immediately after the procedure
  Would the patient recommend the procedure to a friend or family member with the same condition? (5 point Likert scale, 1 = definitely not, 5 = definitely)
Acute procedural success | Immediately after the procedure
  Were all pulmonary veins isolated at procedure end?
Procedure Duration | During procedure
  Skin-to-skin time - i.e. from first needle insertion to withdrawal of sheaths
Fluoroscopy Duration | During procedure
  Time spent with x-ray active
Left atrial dwell time | During procedure
  Time spent with catheters inside the left atrium
Ablation Duration | During procedure
  Time from first ablation application to end of final ablation application
Sedative and anaesthetic drug doses | During procedure
  Doses of sedatives, analgesics and anaesthetics administered during the procedure
Acute Procedural Complications | Immediately after the procedure
  Whether any complications occurred
Same-day discharge rates | 24 hours
  How many patients per arm went home on the same day as their procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Liverpool Heart and Chest Hospital, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Anonymised dataset can be made available upon reasonable request. Identifiable data will not be made available for confidentiality reasons.